CLINICAL TRIAL: NCT01508520
Title: a Prospective Study on the Efficacy of Magnifying Endoscopy With Narrow-band Imaging in Diagnosing Gastric Lesions
Status: Completed | Type: Observational
Sponsor: Xiaobo Li (Other)
Responsible Party: Sponsor-Investigator, Xiaobo Li, Shanghai Institute of Digestive Disease，Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Other Study IDs: rjyyxhk6056
Record Dates: First submitted 2012-01-08; First posted 2012-01-12 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Stomach Neoplasms
Keywords: early gastric cancer; stomach neoplasms; magnifying endoscopy; narrow band imaging
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples after biopsy or resection are to be retained.
Oversight: Data Monitoring Committee: No

SUMMARY:
Magnifying endoscopy with narrow-band imaging (ME-NBI) can emphasize surface pattern and microvascular architecture of the gastric mucosa.However,the usefulness and criteria of NBI for differential diagnosis among early gastric cancers (EGC) have not been fully established.The study is based on the hypothesis:

1. ME-NBI is useful in distinguishing EGC from other gastric lesions
2. ME-NBI is useful in further differential diagnosis among EGCs.

ELIGIBILITY:
Inclusion Criteria:

* patients with gastric lesions which were detected by conventional screening endoscopy and suspected of early malignancy.

Exclusion Criteria:

* advanced gastric cancer or any other malignancy;
* patients under unsuitable conditions for examination or treatment, such as acute upper gastrointestinal bleeding, noncorrectable coagulopathy, severe systemic disease, etc;
* inability to provide informed consent;
* inability to provide histology of resected specimens after endoscopic treatment or surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with gastric lesions suspected of early gastric malignancy
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2009-12; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
diagnosis accuracy of ME-NBI | in 2 weeks after ME-NBI examination
  ME-NBI diagnosis was made during real-time endoscopy procedure and reviewed in two weeks after ME-NBI examination. Sensitivity, specificity, positive predictive value, negative predictive value, and accuracy of ME-NBI diagnosis compared with histology were measured.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaobo Li, MD. Ph.D, Principal Investigator — Shanghai Ren Ji Hospital